CLINICAL TRIAL: NCT07360743
Title: Anti-PD1 Monotherapy in 1L Advanced NSCLC Patients With PD-L1 TPS > 50% and PTI=0
Brief Title: Immunotherapy Without Chemotherapy for Advanced Lung Cancer Patients With High PD-L1 Levels
Acronym: META-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-IMM-2512; 2025-522655-26-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer (Squamous or Non Squamous)
Keywords: anti-PD1 monotherapy; non-small cell lung cancer (NSCLC); Tumor Proportion Score (TPS) >50%; without EGFR/ ALK/ ROS1 mutations; Pro-tumoral inflammatory score (PTI); Advanced metastatic cancers; Personalized immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; cemiplimab

STUDY DESIGN:
Intervention Model Description: META-1 is an academic, open label, multicentric, phase II, proof-of-concept clinical trial designed to evaluate whether a PTI score threshold of 1 could set apart patients at risk of hyperprogression from those who will benefit from long-term anti- PD1 monotherapy while chemotherapy-related toxicities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Anti-PD1 monotherapy in 1L advanced NSCLC patients with PD-L1 TPS > 50% and PTI=0 (Experimental): Pembrolizumab or cemiplimab (anti-PD1) will be considered as investigational medical products (IMP) and will be used in accordance with their marketing authorization for the trial population.
  Interventions: Drug: Pembrolizumab; Drug: Cemiplimab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg every 3 weeks (Q3W) Intravenous (IV) infusion of 30 minutes
  Other Names: KEYTRUDA ®
Drug: Cemiplimab — 350 mg every 3 weeks (Q3W) Intravenous (IV) infusion of 30 minutes
  Other Names: Libtayo®

SUMMARY:
Anti-PD-1 monotherapy has demonstrated significant clinical efficacy in advanced or metastatic non-small cell lung cancer (NSCLC) with high PD-L1 expression (tumor proportion score [TPS] >50%), outperforming platinum-based chemotherapy in terms of objective response rate (ORR) and overall survival (OS). Pivotal randomized trials such as KEYNOTE-024 and EMPOWER-Lung 1 established the superiority of PD-1 blockade in this patient population, leading to regulatory approvals by both the FDA and EMA for first-line treatment. These studies confirmed that a subset of patients can achieve deep and durable responses with immunotherapy alone, highlighting the potential of immune checkpoint inhibition to provide long-term clinical benefit without the toxicities associated with cytotoxic chemotherapy.

Despite these successes, accumulating clinical evidence has revealed a clinically significant risk of hyperprogressive disease (HPD) in a subset of patients treated with anti-PD-1 monotherapy. HPD is characterized by an unexpected and rapid acceleration of tumor growth following treatment initiation and is associated with early clinical deterioration and increased mortality. This phenomenon likely contributes to the early crossover of survival curves frequently observed when comparing immunotherapy alone with chemotherapy in first-line NSCLC trials. In contrast, such early survival crossover is not observed in trials comparing chemotherapy-immunotherapy combinations with chemotherapy alone, including CheckMate-227, CheckMate-9LA, KEYNOTE-189, and KEYNOTE-407. These results have led many thoracic oncologists to favor combined chemo-immunotherapy regimens as first-line treatment, as they reduce the risk of HPD and increase initial ORR.

However, while chemotherapy combined with immunotherapy effectively mitigates the risk of hyperprogression and improves early response rates, it also appears to compromise the durability of antitumor immune responses. Clinical data indicate that the median duration of response with chemo-immunotherapy combinations is approximately 10-11 months, compared with more than 22 months for anti-PD-1 monotherapy alone. This difference is likely attributable to the cytotoxic effects of chemotherapy on immune effector cells, which may limit the persistence and depth of immune-mediated tumor control. Consequently, there remains a strong clinical need to identify patients who could safely and effectively benefit from anti-PD-1 monotherapy while avoiding unnecessary exposure to chemotherapy.

Multiple early-phase translational studies have independently identified soluble plasma biomarkers associated with response or resistance to PD-1 blockade in advanced NSCLC. Building on this body of evidence, translational analyses conducted at Gustave Roussy Cancer Center have identified a composite signature of circulating soluble factors, including interleukin-6 (IL-6), interleukin-8 (IL-8), soluble CD14 (sCD14), soluble CD25 (sCD25), and growth differentiation factor-15 (GDF-15). Together, these biomarkers define a Pro-Tumoral Inflammation (PTI) signature that is strongly associated with primary resistance to anti-PD-1 monotherapy. Elevated PTI scores reflect a systemic inflammatory state that promotes tumor progression and immune dysfunction, and have been linked to poor clinical outcomes, including non-response and hyperprogressive disease.

Within the META-1 sub-protocol of the METAREM master protocol, the investigators propose to integrate these soluble biomarkers into a single PTI score generated through baseline PORTRAIT immunoprofiling. The primary objective of this approach is to prospectively validate the predictive value of the PTI score for anti-PD-1 monotherapy efficacy in advanced NSCLC. By enabling early identification of patients at high risk of resistance or hyperprogression, this strategy aims to refine patient stratification and guide first-line treatment selection. Ultimately, the use of the PTI score could allow clinicians to identify patients most likely to benefit from anti-PD-1 monotherapy, preserving the potential for durable responses while sparing others from ineffective treatment and optimizing the overall therapeutic strategy in advanced NSCLC.

DETAILED DESCRIPTION:
Traditionally, anticancer drug development has been guided by tumor histology and largely focused on tissue-specific characteristics rather than the underlying biological mechanisms driving disease progression. Conventional anticancer therapies, which are often nonspecific, are associated with substantial toxicity and adverse events, and their efficacy frequently diminishes over time due to the emergence of drug resistance. These limitations have driven a paradigm shift toward the development of therapies that target the molecular and biological features of cancer rather than its anatomical origin.

Advances in tumor biology and immunology have profoundly transformed the oncology treatment landscape. Once considered speculative, biomarker-driven and tissue-agnostic therapeutic approaches are now supported by robust clinical evidence. Since 2017, regulatory approvals have validated this shift, beginning with the FDA approval of pembrolizumab for tumors characterized by high microsatellite instability (MSI-H), followed by additional tumor-agnostic agents. To date, seven therapies have received FDA approval for tissue-agnostic indications, underscoring the clinical relevance of shared biological features across cancer types.

A comprehensive understanding of drug mechanisms of action, together with an in-depth assessment of the tumor microenvironment and its inflammatory status, has emerged as a critical determinant of treatment efficacy, particularly in patients who fail to respond to conventional therapies. The increasing focus on immune-tumor interactions has led to the identification of key immune regulatory pathways that represent attractive targets for tumor-agnostic drug development. Among these, CD8⁺ T-cell immunophenotypes play a central role in mediating responses to immunotherapy. Unlike classical oncogenic driver alterations, immune checkpoint molecules such as PD-1 and PD-L1 are not mutated in PD-L1-positive tumors. Nevertheless, PD-L1 expression has been observed across multiple cancer types with otherwise unrelated genomic alterations, making the PD-1/PD-L1 axis a prototypical tumor-agnostic therapeutic target. Pharmacological blockade of this pathway using monoclonal antibodies can restore antitumor T-cell activity and induce meaningful clinical responses.

Anti-PD-1 monotherapy has demonstrated substantial clinical benefit in advanced or metastatic non-small cell lung cancer (NSCLC) with high PD-L1 expression (tumor proportion score [TPS] >50%) across multiple randomized clinical trials. In the KEYNOTE-024 study, pembrolizumab significantly improved objective response rate (ORR) and overall survival (OS) compared with platinum-based chemotherapy. At a median follow-up of 24 months, median OS was 26.3 months for pembrolizumab versus 13.4 months for chemotherapy, with a hazard ratio of 0.62. Notably, the estimated 5-year OS rate was 31.9% in the pembrolizumab arm compared with 16.3% in the chemotherapy arm, highlighting the potential for long-term disease control with immunotherapy.

Similarly, the EMPOWER-Lung 1 trial demonstrated the superiority of cemiplimab over chemotherapy in patients with PD-L1 TPS ≥50%. Median OS was not reached in the cemiplimab arm versus 14.2 months with chemotherapy, and progression-free survival (PFS) was significantly prolonged. Importantly, these benefits were observed despite a high crossover rate, reinforcing the robustness of the survival advantage conferred by PD-1 blockade.

The KEYNOTE-042 study further extended these findings by demonstrating an overall survival benefit for pembrolizumab across PD-L1 TPS subgroups (≥50%, ≥20%, and ≥1%). These results supported the extension of pembrolizumab monotherapy as a first-line option for patients with locally advanced or metastatic NSCLC lacking EGFR or ALK alterations, including those with lower PD-L1 expression levels.

Collectively, these data led to FDA and EMA approvals of anti-PD-1 antibodies, including pembrolizumab and cemiplimab, as first-line monotherapy for advanced or metastatic NSCLC with PD-L1 TPS >50%, as assessed by companion diagnostic immunohistochemistry assays. However, emerging clinical evidence has identified a subset of patients who experience paradoxical hyperprogressive disease (HPD) following initiation of anti-PD-1 monotherapy. HPD is characterized by rapid acceleration of tumor growth and is associated with early mortality. This phenomenon likely explains the early crossover of survival curves observed in trials comparing immunotherapy monotherapy with chemotherapy.

In contrast, such early survival crossover is not observed in studies comparing chemotherapy alone with chemotherapy-immunotherapy combinations, including CheckMate-227, CheckMate-9LA, KEYNOTE-189, and KEYNOTE-407. As a result, many thoracic oncologists, particularly in France, have adopted chemo-immunotherapy combinations as first-line treatment for PD-L1-high NSCLC, as these regimens increase ORR and reduce the risk of hyperprogression. However, this approach exposes patients who would otherwise benefit from anti-PD-1 monotherapy-estimated at approximately 40% of PD-L1-high NSCLC cases-to unnecessary chemotherapy-related toxicity, potentially compromising long-term survival and quality of life.

Supporting this concern, a recent systematic review and reconstructed individual patient data analysis examined the impact of platinum-based chemotherapy (PCT) combined with immune checkpoint inhibitors in metastatic NSCLC. This analysis demonstrated that PCT-containing regimens were associated with a higher risk of acquired resistance at 12 months and a shorter median duration of response compared with PCT-free immunotherapy combinations. In contrast, the addition of CTLA-4 inhibitors did not significantly increase resistance rates. These findings suggest that while chemotherapy may enhance early disease control, it may also accelerate the development of resistance to immune checkpoint blockade.

Taken together, these observations emphasize the urgent need to refine patient selection and optimize treatment sequencing in NSCLC immunotherapy. Multiple early-phase studies have independently identified soluble plasma biomarkers with predictive value for anti-PD-1 monotherapy efficacy. Building on this work, translational analyses conducted at Gustave Roussy Cancer Center identified a composite signature of circulating soluble biomarkers-including interleukin-6 (IL-6), interleukin-8 (IL-8), soluble CD14 (sCD14), soluble CD25 (sCD25), and growth differentiation factor-15 (GDF-15). This Pro-Tumoral Inflammation (PTI) signature is strongly associated with primary resistance to anti-PD-1 therapy and provides a biologically grounded framework for improving patient stratification and therapeutic decision-making in advanced NSCLC. depending on their PTI score, some patients could be identified early on as being at higher risk of non-response (including hyperprogression) under anti-PD1 monotherapy.

Here the investigators aim to implement those biomarkers in an exploratory sub-protocol of the METAREM master protocol for a prospective validation of their value to stratify NSCLC patient's care.

Thus, META-1 trial aims to incorporate PTI score as a biomarker for patient selection via baseline PORTRAIT profile. In the REMISSION program, which includes METAREM master protocol and its sub-protocols, the Meso Scale Discovery multiplex ultrasensitive titration platform will be used to titrate the cytokine levels in plasma from NSCLC patients which will permit to establish the PTI score for patient selection.

META-1 is a prospective, French, multicentric, phase II, sub-protocol of the METAREM master protocol. META-1 focuses on evaluating the value of the PTI score to identify patients who could benefit from the long-term efficacy an anti-PD1 monotherapy, while avoiding the risk of hyperprogression and the toxicities of chemotherapy. Using ultrasensitive methods, the patient's plasma samples (collected for baseline PORTRAIT) will be rapidly analysed. Based on PTI score cut-off levels i.e., patients with PTI=0, the patient will be selected for inclusion in the META-1 trial.

Designed as an academic proof-of-concept study, META-1 aims to validate the hypothesis that can enable personalized benefit-risk predictions, helping identify the most advantageous treatment for advanced NSCLC patients.

Of note, both anti-PD1 monotherapy and anti-PD1 in combination with carboplatin doublet chemotherapies are currently standard of care options as first-line treatment for advanced NSCLC with PD-L1 TPS > 50%. The choice of one or the other treatment option currently relies on the sole practitioner choice without objective decision criteria.

Trial aim to demonstrate that blood titration of the PTI score can help to orient patients to one or the other treatment option with a biological rationale and an objective titration of soluble blood factors.

META-1 trial involves the following key steps:

Patient selection will be based on the eligibility and inclusion criteria of the METAREM master protocol and the META-1 trial. Only patients who have consented to both the master protocol and the trial are eligible to be included in the META-1 trial. Along with the PORTRAIT immune profile, inclusion criteria are also based on pathology, imaging, clinical setting, and routine biological criteria.

Patients with tumors having a PD-L1 TPS > 50% according to approved CDx IHC assays (using the anti-PD-L1 IHC staining clones 22C3, 28-8 and SP263)11 will be tested at baseline within the PORTRAIT immune profiling.

Fresh blood samples will be mandatory for PORTRAIT analysis prior to inclusion in the META-1 trial, while fresh tumor samples will be optional according to the following scenarios:

1. if patients have already undergone their diagnostic tumor biopsy to establish their PD-L1 IHC score before signing the METAREM master protocol consent, a new baseline PORTRAIT tumor biopsy will be optional. Archived diagnostic tumor samples may be used.
2. if patients provide consent for the METAREM prior to their initial diagnostic tumor biopsy, the baseline PORTRAIT analysis may be performed on that fresh tumor biopsy.
3. A minimum of 10 FFPE blank slides should be made available at baseline either from a previous tumor biopsy or a new one performed during the METAREM screening period. If no baseline tumor material is available and a new tumor biopsy cannot be performed, the investigator must request an exemption from the tumor biopsy requirement from both the sponsor and the coordinating investigator of the META-1 trial.

   1. Patients with PTI score = zero - low levels of IL6, IL8, sCD14, sCD25 and GDF15 - will be eligible to participate in the META-1 trial and receive anti-PD1 monotherapy (pembrolizumab or cemiplimab) according to the approved and reimbursed standard of care (SoC) in France.

      Once enrolled into the META-1 trial, patients will be treated with an anti-PD1 monotherapy per standard of care (pembrolizumab or cemiplimab) until disease progression, unacceptable toxicity, death, investigator's decision, or patient's decision.

      For patients whose initial baseline tumor biopsy for PORTRAIT has been collected, an on-treatment PORTRAIT analysis will be repeated at C2D1 (W3) for immune profiling. As with the baseline biopsy, the on-treatment tumor biopsy will not be mandatory, as patients will be treated according to the standard of care.

      RECIST v1.1 imaging assessment should be performed by the investigator at the screening visit (baseline PORTRAIT), the inclusion visit, C3D1 (W6) and C5D1 (W12) according to the SoC. After 12 weeks of treatment, subsequent RECIST v1.1 imaging assessment should be performed by the investigator as per the SoC schedule and local site practices during treatment and follow-up period, until documented disease progression or death, whichever occurs first, for a maximum follow-up period of 36 months.
   2. Patients with PTI score ≥ 1 - high levels of IL6, IL8, sCD14, sCD25 and GDF15 - will be followed for up to 36 months according to the SoC to assess disease progression and overall survival, provided they have given their consent. Throughout the study, radiological examinations and tumor assessments by the investigator will be performed in accordance with the SoC. Patients will receive standard treatment at the discretion of the treating physician. Information on treatments and any newly initiated therapies will also be collected. These patients will not undergo any sampling during the META-1 trial, except for samples collected during the screening visit conducted under the METAREM master protocol.

ELIGIBILITY:
Inclusion Criteria:

In addition to the inclusion criteria of the METAREM master protocol, following additional criteria must be respected during patient inclusion in META-1 trial:

1. Patients with age ≥18 years
2. Patients in first-line therapy for advanced metastatic NSCLC with PD-L1 Tumor Proportion Score (TPS) >50%, without EGFR/ ALK/ ROS1 mutations and irrespective of their histological subtype (squamous or non-squamous).
3. Patients with a PTI score of zero in plasma on the baseline PORTRAIT report. Note: Patients with PTI score ≥ 1 who meet all other criteria will be followed up to 36 months or death according to standard of care.

Exclusion Criteria:

In addition to the Exclusion criteria of the METAREM master protocol, following additional criteria must be considered during patient exclusion from META-1 trial:

1. Patients who have previously received an anti-PD(L)1 or anti-CTLA4 or anti-LAG-3 or anti-TIM3 immunotherapy.
2. Patients with any Hypersensitivity to the active ingredient or to any of the excipients of Pembrolizumab or Cemiplimab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the rate of patients without early progression upon anti-PD1 monotherapy by selecting patients with a baseline plasma PTI score of 0 in patients with advanced/metastatic NSCLC with PD-L1 TPS >50%. | 12 weeks
  The primary endpoint is the rate of patients without disease progression at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David PLANCHARD, MD, PHD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris